CLINICAL TRIAL: NCT05894395
Title: A Cross-Sectional and Open Pre-Post Interventional Study Evaluating Circulating and Mucosal Humoral and Cell-Mediated Immunity Following Measles, Mumps and Rubella (MMR) Vaccination in Adults
Brief Title: Immunity in Persons Fully Vaccinated Against Measles, Mumps and Rubella and Responses to Booster Vaccination
Acronym: MIPS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MIPS101124
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Mumps; Measles; Rubella
MeSH Terms: conditions — Mumps; Measles; Rubella

STUDY DESIGN:
Intervention Model Description: Participants with two previous lifetime doses of MMR-containing vaccine will be randomized to receive a single M-M-R-VaxPro booster vaccination (3rd lifetime MMR-containing vaccine dose) or no intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MMR Booster Vaccination Arm (Experimental): Participants (adults 18+ having previously received 2 lifetime doses of MMR-containing vaccine) will receive a single MMR booster vaccination (3rd lifetime dose) as M-M-R-VaxPro.
  Interventions: Biological: MMR booster vaccination (as M-M-R-VaxPro)
- Observational Arm (No Intervention): Participants (adults 18+ having previously received 2 lifetime doses of MMR-containing vaccine) will be assessed at study enrollment and at a 1 year follow-up visit

INTERVENTIONS:
Biological: MMR booster vaccination (as M-M-R-VaxPro) — a single dose of MMR-containing vaccine (as M-M-R-VaxPro), in adults having previously received 2 lifetime doses of MMR-containing vaccine
  Arms: MMR Booster Vaccination Arm

SUMMARY:
The purpose of this study is to investigate the immunity of persons fully vaccinated against measles, mumps and rubella and to examine the course of immunity after booster vaccination.

DETAILED DESCRIPTION:
Determining whether individuals respond to vaccination is an important healthcare question with significant public health impact. In recent years there have been surges in cases of measles and mumps; vaccine-preventable diseases which have previously been well-controlled since the introduction of regular vaccination (as MMR) in the 1970s-80s. Since 2016, approximately 10,000-15,000 cases each of measles and mumps have been reported annually in Europe. Despite high vaccination coverage and being declared "measles endemic free", multiple outbreaks have occurred in Switzerland, affecting predominately older adults and young children. While rubella cases remain relatively uncommon, infection during pregnancy can result in Congenital Rubella Syndrome and lead to severe birth defects, underscoring the importance of adequate prevention. All three viruses are highly contagious and transmitted through the oral/respiratory mucosal tissue by contact with infected respiratory secretions.

Importantly, in recent years approximately 30% of measles cases and up to half of mumps cases have been found to occur in individuals receiving at least 2 previous MMR doses, suggesting waning immunity. Although seroconversion after two doses of mumps vaccine (as MMR) nears 90-100%, field effectiveness is closer to 88% (range 75-95%). Booster immunization, however, is not currently indicated in adults. Furthermore, while serum virus-neutralizing antibodies are evaluated as an indicator of responsiveness following mumps vaccination, they are not the correlate of protective immunity. There is need to better understand both 1) The duration of vaccine-elicited protection to all three viruses; and 2) The underlying protective immune mechanisms elicited by vaccination.

Assessments of vaccine responses most often utilize blood to evaluate the establishment of circulating immunity, typically antibodies, in individuals. While antibody responses may predict response to vaccination they may or may not be the immune subset actually responsible for protection. Furthermore, circulating immune responses detectable in the blood are not necessarily representative of responses occurring at mucosal sites. Samples such as saliva, sputum or nasal washes, in contrast, can be collected with relative ease, and can provide insights into the oral and respiratory mucosal environments, which are primary sites of pathogen exposure. Understanding whether specific vaccines elicit immune responses at mucosal sites, that are detectable using minimally-invasive techniques, that correlate with protection from disease, or that can act as a surrogate for circulating responses, would be highly valuable in immune monitoring.

With this study the investigators plan to evaluate persisting measles, mumps and rubella seropositivity in previously-vaccinated adults and to assess whether anti-viral immune responses are detectable in saliva (representative of the oral mucosa) as well as how these compare to circulating responses detectable in the blood. In a random subset of study participants they will offer a booster immunization and subsequently evaluate mucosal and circulating immune responses in the saliva, nasal washes (representative of the oral and respiratory mucosae) and blood 7 and 28 days and 1 year post-vaccination to determine whether additional predictive indicators for measles, mumps and/or rubella immunity can be identified.

Significantly, the proposed study has the potential to 1) Provide unique insights into similarities and differences between mucosal and circulating anti-viral immune responses to MMR vaccination as well as the duration of such responses; 2) Aid in the identification of a correlate of immune protection or novel indicator of responsiveness to mumps (and possibly measles and rubella) vaccination; and 3) Improve immune monitoring after MMR vaccination by using saliva and/or nasal washes to reduce invasiveness and provide a proof-of-concept for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-49 (inclusive) at the time of the study screening visit
* Has received exactly two previous doses of MMR-containing vaccine at any point up to one calendar year prior to the study screening visit
* Willing to receive a booster MMR vaccination as outlined in the study protocol
* Able and willing to comply with all other study requirements (attend all study visits and provide blood, saliva, nasal wash samples at each visit as outlined)
* Sufficient language (German or English) and cognitive skills
* Provides written, informed consent to participate in the study

Exclusion Criteria:

* Acute respiratory or other infections (postpone baseline visit until resolved)
* Receipt of any other vaccination less than 4 weeks prior to the baseline visit or intention to receive another vaccination within 4 weeks following the baseline visit
* Previous hypersensitivity reaction following receipt of any MMR-containing vaccine or previous hypersensitivity reaction to any component of M-M-R-vaxPro
* Pregnancy, lactation, or intention to become pregnant during the study
* Individuals with confirmed or suspected immunosuppressive or immune-deficient state
* Known current or chronic or severe disease
* Receipt of blood or plasma transfusions, or administration of immune globulin (IG) less than 12 weeks prior to the baseline visit, or intention to receive IG within 4 weeks following the baseline visit
* Any other significant disease, disorder, or finding which could potentially result in an increased risk to the volunteer due to participation in the study
* Being enrolled in another interventional study that may interfere with the current study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity post MMR-booster vaccination | From admission to one year post vaccination
  Immunogenicity will be assessed by evaluating anti-measles, -mumps, and -rubella serum Immunoglobulin G (IgG) titers post-booster vaccination. A 5-fold increase in titers for each virus between baseline (day 0) and day 28 post-booster vaccination will be considered "immunogenic".

SECONDARY OUTCOMES:
Assessment of Immunoglobulin A (IgA) blood and mucosal immune responses to each virus (measles, mumps, and rubella) | From admission to one year post vaccination
  From screened participants, population-level IgA responses to measles, mumps, and rubella will be estimated. Virus-specific IgA responses in serum, saliva and nasal washes will be assessed at each timepoint by Enzyme-Linked Immunosorbent Assay (ELISA) and compared over time (day 0/ day 7/ day 28/ 1 year).
Assessment of Immunoglobulin G (IgG) blood and mucosal immune responses to each virus (measles, mumps, and rubella) | From admission to one year post vaccination
  From screened participants, population-level IgG responses to measles, mumps, and rubella will be estimated. Virus-specific IgG responses in serum, saliva and nasal washes will be assessed at each timepoint by Enzyme-Linked Fluorescent Assay (ELFA) and compared over time (day 0/ day 7/ day 28/ 1 year).
Assessment of virus-specific B cell blood and mucosal immune responses to each virus (measles, mumps, and rubella) | From admission to one year post vaccination
  From screened participants, population-level virus-specific B cell responses to measles, mumps, and rubella will be estimated. Virus-specific B cell responses in blood, saliva and nasal washes will be assessed at each timepoint by IgG Enzyme-Linked Immunosorbent Spot (ELISpot) assay and compared over time (day 0/ day 7/ day 28/ 1 year).
Assessment of virus-specific T cell blood and mucosal immune responses to each virus (measles, mumps, and rubella) | From admission to one year post vaccination
  From screened participants, population-level virus-specific T cell responses to measles, mumps, and rubella will be estimated. Virus-specific T cell responses in blood, saliva and nasal washes will be assessed at each timepoint by Interferon-gamma (IFN-gamma) ELISpot assay and compared over time (day 0/ day 7/ day 28/ 1 year).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Fehr, M.D., Principal Investigator — Department Head
Locations (1):
- Epidemiology, Biostatistics and Prevention Institute University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No